CLINICAL TRIAL: NCT06321835
Title: The Effect of Different Patient Positions on Endotracheal Tube Cuff Pressure in Patients Undergoing Urological Procedures: A Prospective Study
Brief Title: The Effect of Different Patient Positions on Endotracheal Tube Cuff Pressure
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nursen Karaca, Medical Doctor, Ege University
Other Study IDs: 16-10/13
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Endotracheal Tube Cuff Pressure; Patient Positions
Keywords: endotracheal tube; cuff pressure; patient position; prone; lateral flank; litotomy; sore throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Supine Group: The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy.
  Interventions: Procedure: Endotracheal tube cuff pressure measurement
- Prone Group: The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy.
  Interventions: Procedure: Endotracheal tube cuff pressure measurement
- Lithotomy Group: The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy.
  Interventions: Procedure: Endotracheal tube cuff pressure measurement
- Lateral flank group: The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy.
  Interventions: Procedure: Endotracheal tube cuff pressure measurement

INTERVENTIONS:
Procedure: Endotracheal tube cuff pressure measurement — This is a prospective study conducted on 200 patients undergoing urological procedures in supine, prone, lateral flank and litotomy positions. After intubation (T0), the cuff pressure was checked with a cuff manometer and adjusted at 25 cmH2O as the baseline and continuously monitored. The cuff pressure was checked again before (T1) and after achieving the final position (T2) and then at 5 (T3), 10 (T4), 15 (T5), 30, 45, 60, 90, 120, 150, 180 minutes after the position, at the end of the procedure (T6) and before extubation (T7). At postoperative 2nd and 12th hours, the patients were interviewed for sore throat, hoarseness and cough.

SUMMARY:
Background: The placement of a cuffed endotracheal tube for the administration of general anesthesia is a routine procedure. In the part of the intubation tube located in the trachea, there is a balloon (cuff) to prevent gase leakage, aspiration of secretions and gastric contents into the lungs. Inadequate inflation of cuff may lead to inadequate ventilation, aspiration and associated complications, while excessive inflation may cause complications in ranging from postoperative pharyngeal complaints to tracheal rupture due to increased cuff pressure. This study aimed to determine the effect of different patient positions on the endotracheal cuff pressure in patients undergoing urological procedures.

Methods: This is a prospective study conducted on 200 patients undergoing urological procedures in supine, prone, lateral flank and litotomy positions. After intubation (T0), the cuff pressure was checked with a cuff manometer and adjusted at 25 cmH2O as the baseline and continuously monitored. The cuff pressure was checked again before (T1) and after achieving the final position (T2) and then at 5 (T3), 10 (T4), 15 (T5), 30, 45, 60, 90, 120, 150, 180 minutes after the position, at the end of the procedure (T6) and before extubation (T7). At postoperative 2nd and 12th hours, the patients were interviewed for sore throat, hoarseness and cough.

DETAILED DESCRIPTION:
After Institutional Review Board approval from Ege University (Ethical Committee No. 16-10/13, 09.12.2016) and written informed consent, 200 patients aged 18-75 years, ASA physical status I-II, who were planned for elective urological surgery in one of the supine, prone, lateral flank or lithotomy position were studied. The exclusion criteria were as follows: emergency operation, a history of chronic lung disease, upper and/or lower respiratory tract infection within 2 weeks before surgery, morbid obesity, pregnancy, laparoscopic surgery, single lung ventilation, difficut airway, hemodynamic instability and/or respiratory complications in the intraoperative period, history of mental illness or communication problems.

The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy. After the patient was taken to the operating room, routine vital sign monitoring of non-invasive arterial blood pressure (NIBP), electrocardiogram (ECG) and pulse oximetry (SpO2) was performed. Oxygen mask was connected and 3 minutes %100 preoxygenation was applied. Intravenous (IV) vascular access was provided and fluid therapy was started. For induction of general anesthesia, 10 mcg/kg atropine, 1mg/kg lidocaine, 2-3 mg/kg propofol, 1-3 µg/kg fentanyl and 0,6 mg/kg rocuronium bromide were administered intravenously.

After adequate mask ventilation, female patients were intubated orotracheally with a tube of internal diameter (ID) 7-7.5mm, while male patients were intubated with a tube of ID 8-8.5mm. The equal ventilation of both lungs was confirmed by oscultation, and the position of the endotracheal tube was determined after observing the waveform of ETCO2 on the capnograph. High volume, low pressure endotracheal tubes were used for intubation. Patients who were to undergo surgery in the prone position were also intubated with a spiral tube of the same number. After intubation, the cuff of the ETT was inflated with air through an injector of 5-10 mL as a standard method, and the pressure value of the cuff after intubation (T0) was measured and recorded in a neutral head position using an analog cuff manometer (VBM Medizintechnik®, GmbH, Germany). Immediately after that, the cuff pressure was adjusted to 25 cmH2O. The manometer continuously monitored the cuff pressure without separating it from the pilot balloon of the ETT. The patient was taken volume-controlled mechanical ventilation support with a tidal volume of 6-8 mL/kg, respiratory rate of 12-16/min, and ETCO2 of 35-40 mmHg. For anesthesia maintenance, a mixture of 50% O2 and air was used, along with Sevoflurane (Sevorane Liquid 250 ml®, Abbott, UK) at 2% MAC and remifentanil infusion.

Before and after giving the patient the necessary position for the operation, the cuff pressure was measured and recorded at T1 and T2, respectively. After giving the position, attention was paid to keeping the head in a neutral position relative to the body. To prevent the effect of airway pressure on the manometer during cuff pressure measurement, the value seen at the end of expiration was recorded. Subsequently, values at 5 minutes (T3), 10 minutes (T4), 15 minutes (T5), 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, and 180 minutes were recorded during the operation. In addition, during the operation, parameters such as blood pressure, heart rate, SpO2, end-tidal CO2 (ETCO2), tidal volume, respiratory rate, mean airway pressure (MAP), and peak airway pressure (PAP) were monitored and recorded. There was no intervention in cuff pressure values during the monitoring period. Finally, after the surgical procedure was completed (T6) and before extubation after patients were put in a neutral (supine) position for waking up, cuff pressure and other parameter values were recorded. Patients were interviewed to determine if they had any complaints of sore throat, hoarseness, or cough at postoperative 2nd and 12th hours.

According to a previous study (10) the mean (SD) ETT cuff pressure was increased by 6.5 (3.9) cm H2O after the positional change from the supine to the lateral decubitus position. Assuming that the difference in the mean cuff pressure is reduced by 50% (3.25 cm H2O), we calculated that 23 patients would be needed in each group with a = 0.05 and b = 0.20. In our study, 50 patients per group were included.

The data were analyzed using the SPSS for Windows 21.0 software. Demographic data were calculated as mean standart deviation (min-max). Differences between data were analyzed using the t-test. For comparing repeated measurements, One-Way Analysis of Variance (One-Way ANOVA) was used. Post Hoc tests were used for between group comparisons. A p-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 200 patients aged 18-75 years
* ASA physical status I-II
* Who were planned for elective urological surgery in one of the supine, prone, lateral flank or lithotomy position were studied

Exclusion Criteria:

* emergency operation
* a history of chronic lung disease
* upper and/or lower respiratory tract infection within 2 weeks before surgery
* morbid obesity
* pregnancy
* laparoscopic surgery
* single lung ventilation
* difficut airway
* hemodynamic instability and/or respiratory complications in the intraoperative period
* history of mental illness or communication problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients aged 18-75 years, ASA physical status I-II, who were planned for elective urological surgery in one of the supine, prone, lateral flank or lithotomy position were studied. The patients were divided into four groups according to the operation position as supine, lateral flank, prone and lithotomy
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
The Effect of Different Patient Positions on Endotracheal Tube Cuff Pressure in Patients Undergoing Urological Procedures: A Prospective Study | 1 year
  Primary outcome of this study is endotracheal cuff pressure can be changed in patients undergoing urological procedures in different patient positions.

SECONDARY OUTCOMES:
The Effect of Different Patient Positions on Endotracheal Tube Cuff Pressure in Patients | 1 year
  Secondary outcome of this study is the change of endotracheal cuff pressure can have effect on the postoperative pharyngolaryngeal complications

IPD SHARING:
Plan to Share IPD: No